CLINICAL TRIAL: NCT04448132
Title: Evaluation of the Persistence of the Immunity in 4-year-old Children Previously Immunised With an Adjuvanted Reduced Dose Inactivated Polio Vaccine, IPV-Al AJV (Picovax®) by Measuring the Response to an Additional Dose of IPV-Al AJV
Brief Title: Evaluation of Persistence of Immunity in 4-year-old Children Previously Immunised With IPV-Al AJV (Picovax®)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AJ Vaccines A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VIPV-07 E2
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPV-Al AJV (Experimental): One dose of 0.5 mL of IPV-Al AJV injected intramuscularly perpendicular to the skin in the RIGHT deltoid muscle.
  Interventions: Biological: IPV-Al

INTERVENTIONS:
Biological: IPV-Al — adjuvanted reduced dose inactivated polio vaccine
  Other Names: Picovax®; IPV-Al AJV

SUMMARY:
The trial is a phase 4, open-label, multicentre clinical trial with healthy subjects who have been vaccinated with IPV-Al AJV at 2, 4, 6 and 15 18 months of age in previous trials. Levels of antibodies against poliovirus types 1, 2 and 3 after immunisation with IPV Al AJV will be measured in the trial subjects at the age of 4 years. An additional IPV-Al AJV dose (investigational vaccine) will be administered and the booster response to IPV-Al AJV will be investigated one month after administration.

ELIGIBILITY:
Inclusion Criteria:

1. Children that have been vaccinated with IPV-Al AJV in the VIPV-07 and VIPV-07 E1 trials and have completed these trials
2. Healthy, as assessed from medical history and physical examination
3. Parent(s)/guardian(s), according to the local legal requirements, have been properly informed about the trial and have signed the informed consent form
4. Parent(s)/guardian(s), according to the local legal requirements, have been granted access to the child´s trial related medical records
5. Parent(s)/guardian(s), according to the local legal requirements, are likely to comply with trial procedures

Exclusion Criteria:

1. Previous vaccination with OPV
2. Previous vaccination with IPV outside the VIPV-07 and VIPV-07 E1 trials
3. Known or suspected immunodeficiency (e.g. leukaemia, lymphoma) or family history of congenital or hereditary immunodeficiency. HIV is not an exclusion criterion.
4. Severe uncontrolled chronic (e.g. neurologic, pulmonary, gastrointestinal, hepatic, renal or endocrine) disease
5. Known or suspected allergy to vaccine constituents (e.g. hypersensitivity to formaldehyde and/or 2-phenoxy-ethanol)
6. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections or blood sampling
7. Treatment with a product which is likely to modify the immune response (e.g. blood products and immunoglobulins) prior to inclusion or planned during the trial period
8. Participating in another interventional clinical trial
9. Not suitable for inclusion in the opinion of the investigator

Ages: 4 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Seroprotection (titer ≥8) against poliovirus types 1, 2 and 3 | One month after administration of an additional dose of IPV-Al AJV
  Individual serum titers against poliovirus types 1, 2 and three will be measured in collected serum samples

CONTACTS AND LOCATIONS:
Locations (1):
- Cevaxim, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saez-Llorens X, Chan M, DeAntonio R, Petersen T, Olesen C, Jensen JS, Sorensen C, Ekstrand LM, Czort MK, Kristensen HH, Thulstrup N, Christoffersen DB. Persistence of protective anti-poliovirus antibody levels in 4-year-old children previously primed with Picovax(R), a trivalent, aluminium-adjuvanted reduced dose inactivated polio vaccine. Vaccine. 2022 Sep 22;40(40):5835-5841. doi: 10.1016/j.vaccine.2022.06.084. Epub 2022 Sep 3. PMID 36064670